CLINICAL TRIAL: NCT04336241
Title: An Open-Label, Multicenter, Phase 1 Study of RP2 as a Single Agent and in Combination With PD1 Blockade in Patients With Solid Tumors
Brief Title: Study of RP2 Monotherapy and RP2 in Combination With Nivolumab in Patients With Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Replimune Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RP2-001-18
Record Dates: First submitted 2020-03-17; First posted 2020-04-07 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Cancer
Keywords: Uveal Melanoma; Gastrointestinal Cancers; Lung Cancer; Breast Cancer
MeSH Terms: conditions — Neoplasms; Uveal Melanoma; Gastrointestinal Neoplasms; Lung Neoplasms; Breast Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Part 1 - Dose Escalation - Patients will be enrolled into three sequential dose level cohorts.
  Part 2 - Dose expansion - Patients will receive a fixed dose of RP2 in combination with Nivolumab.
  Part 3 - Patients will receive four doses of RP2 monotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Dose escalation of RP2 - superficial tumors (Experimental): Dose escalation of RP2 alone in 3 cohorts with IT injections in superficial tumors.
  Interventions: Biological: RP2
- Dose escalation of RP2 - deep/visceral tumors (Experimental): Dose escalation of RP2 alone in 3 cohorts with imaging guided IT injections in deep/visceral tumors.
  Interventions: Biological: RP2
- Dose expansion of RP2 and nivolumab - superficial tumors (Experimental): Doses of RP2 (IT) in superficial tumors with nivolumab (IV).
  Interventions: Biological: RP2; Biological: nivolumab
- Dose expansion of RP2 and nivolumab - deep/visceral tumors (Experimental): Imaging guided doses of RP2 (IT) in deep/visceral tumors.
  Interventions: Biological: RP2; Biological: nivolumab
- Seronegative cohort (Experimental): Doses of RP2 (IT) in HSV seronegative participants.
  Interventions: Biological: RP2

INTERVENTIONS:
Biological: RP2 — Genetically modified herpes simplex type 1 virus for tumor lysis and immune stimulation
Biological: nivolumab — Programmed death receptor (PD-1) blocking antibody
  Other Names: Opdivo
  Arms: Dose expansion of RP2 and nivolumab - deep/visceral tumors; Dose expansion of RP2 and nivolumab - superficial tumors

SUMMARY:
RP2-001-18 is a Phase 1, multicenter, open label, single agent dose escalation and combination treatment study of RP2 in adult subjects with advanced solid tumors, to determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D), as well as to evaluate preliminary efficacy.

DETAILED DESCRIPTION:
RP2 is a genetically modified herpes simplex type 1 virus (HSV-1) that expresses an anti-CTLA-4 antibody and is designed to directly destroy tumors and to generate an anti-tumor immune response. This is a Phase 1, multicenter, open label, dose escalation and expansion, first-in-human (FIH) clinical study to evaluate the safety and tolerability, biodistribution, shedding, and preliminary efficacy of RP2 alone and in combination with nivolumab in adult subjects with advanced solid tumors.

The study will be conducted in two parts. The first part of the study is an open-label, dose escalation FIH Phase 1 study to assess the safety and tolerability of RP2 and to determine the recommended Phase 2 dose (RP2D) to be used in the second part of the study. The second part of the study is an open label design to further investigate safety of RP2 in combination with nivolumab. It will also assess the biological activity of multiple doses of RP2 in combination with nivolumab. An expansion to the second part of the study will include enrolment of a further 30 patients on RP2 in combination with nivolumab.

Following completion of the expansion in part 2, part 3 will enroll a further 15 patients on RP3 monotherapy.

The expansion to part 2 and part 3 will focus on patients with advanced or metastatic uveal melanoma, lung cancer, breast cancer or GI cancers and patients with liver metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to participate and comply with all trial requirements and able to provide signed and dated informed consent prior to initiation of any trial procedures
* Male or Female ≥ 18 years of age
* Patients with advanced or metastatic non-neurological solid tumors, who have progressed on standard therapy or cannot tolerate standard therapy, or for which there is no standard therapy preferred to enrolment in a clinical trial
* Consent to provide archival tumour biopsy samples within 6 months, or a fresh tumour biopsy is needed. Patients must also consent to provide on-treatment biopsies as per protocol
* At least one measurable and injectable tumor of ≥ 1 cm in longest diameter (or shorter diameter for lymph nodes).
* Women of child-bearing potential (WOCBP) must have a negative urine pregnancy test at screening and a negative urine pregnancy test prior to administration of each dose of RP2 or nivolumab
* WOCBP must agree to use adequate birth control throughout their participation and for 3 months after RP2 alone and 5 months after nivolumab last study treatment
* Males with partners of child-bearing potential must agree to use adequate birth control throughout their participation and for 3 months for RP2 alone and 7 months after nivolumab last study treatment
* Have laboratory values (obtained ≤ 28 days prior to first infusion day) in accordance with the study protocol
* Have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1

Cohort 2a only:

* Baseline ECG that does not show abnormalities according to the protocol
* Baseline troponin < 0.06 ng/mL
* Baseline oxygen saturation levels that do not show abnormalities according to the protocol

Cohort 2b and Part 3 only:

* Patients in Cohort 2b should have histologically or cytologically confirmed diagnosis of advanced or metastatic uveal melanoma, lung cancer, breast cancer, or gastrointestinal cancers (including but not limited to colorectal cancer [CRC] [microsatellite stable], gastric cancer, gastroesophageal junction cancer, and oesophageal cancer) (n=30)
* Patients with HCC and a diagnosis of hepatitis B must be off antiviral therapy for at least 4 weeks prior to enrollment.
* Patients with acute or chronic hepatitis B or C must be expected to not require antiviral therapy during the RP2 treatment period.
* Patients with HCC who have evidence of acute or chronic hepatitis C infection must have completed treatment for hepatitis C at least 1 month prior to study enrollment
* Patients in Part 3 should have solid tumours (excluding skin cancers) that the investigator deems suitable for RP2 monotherapy, including at least 10 patients with liver metastases from prevalent tumour types (e.g. lung, breast [including recurrent chest wall], and gastrointestinal cancers [colorectal, gastric, and oesophageal cancers]) (n=15)
* Patient has progressed during or after one to three prior systemic anticancer therapies for advanced or metastatic disease or during or within six months of receiving adjuvant therapy. Patients who, in the opinion of the investigator, are deemed not appropriate candidates for standard-of-care systemic anticancer therapy for advanced or metastatic disease, or who, after documented consultation with their treating physician, refuse standard-of-care systemic anticancer therapy may be eligible after discussion with the medical monitor

Exclusion Criteria:

* Prior treatment with an oncolytic virus therapy
* History of viral infections according to the protocol
* Systemic infection requiring IV antibiotics within 14 days prior to dosing
* Prior complications with herpes infections
* Chronic use of anti-virals
* Systemic therapies for cancer within five half-lives or 4 weeks of first dose; whichever is shorter
* Conditions that require certain doses of steroids (some doses and types will be permitted)
* Known active brain metastases - previously treated brain metastases may be permitted
* Major surgery ≤ 2 weeks prior to starting study drug
* Prior malignancy active with the previous 3 years; except for locally curable cancers that have apparently been cured
* Female who has a positive urine pregnancy test or is breast-feeding or planning to become pregnant during study treatment and 90 days for RP2 alone or 5 months for RP2 and nivolumab after the last dose of treatment
* Participation in another clinical study within 4 weeks prior to the first dose
* History of myocarditis or congestive heart failure (as defined by the New York Heart Association Functional Classification III or IV), or unstable angina, serious uncontrolled cardiac arrhythmia, uncontrolled infection, or myocardial infarction within 6 months of randomization

  * History of allergy or sensitivity to study drug components
  * Has known psychiatric or substance abuse disorders that would interfere with cooperating with the requirements of the study

Part 2 patients only:

* Participants with history of life-threatening toxicity related to prior immune therapy except those that are likely to re-occur with standard countermeasures
* Treatment with botanical preparations within 2 weeks prior to treatment
* Certain autoimmune diseases, some types will be permitted
* History of interstitial lung disease
* Severe hypersensitivity to another monoclonal antibody
* Has received radiotherapy within 2 weeks of start of study treatment
* Has received a live vaccine within 28 days prior to first dose of study drug
* History of non-infectious pneumonitis
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study
* Other serious or uncontrolled medical disorders

Cohort 2b and Part 3 (only for the subset of patients with liver metastases suitable and intended for injection)

* Presence of liver metastases that are estimated to invade more than one-third of the liver
* Macroscopic intravascular invasion into the main portal vein, hepatic vein or vena cava
* Significant bleeding event within the last 12 months that places the patient at risk for intrahepatic intratumoral injection procedure based on investigator assessment
* Prior chemoembolization, radioembolization, or other locoregional liver-directed procedures to the lesion selected for intratumoral injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-10-17 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of adverse events (AEs) | From Day 1 up to 60 days after last dose
  Percentage of subjects with AEs
Percentage of serious adverse events (SAEs) | From Day 1 up to 60 days after last dose
  Percentage of subjects with SAEs
Percentage of dose limiting toxicities (DLTs) | From Day 1 up to 30 days after last dose.
  Percentage of subjects with DLTs
Percentage of treatment emergent adverse events (TEAEs) | From Day 1 up to 60 days after last dose.
  Percentage of subjects with TEAEs
Percentage of TEAEs ≥ Grade 3 | From Day 1 up to 60 days after last dose.
  Percentage of subjects with TEAEs ≥ Grade 3
Percentage of events requiring withdrawal | From Day 1 up to last dose (up to 8 weeks for dose escalation phase and up to 2 years for expansion phase)).
  Percentage of subjects experiencing events requiring withdrawal from treatment.
Maximum tolerated dose (MTD) of RP2 | 7 months
  MTD on the safety and response data collected during the dose escalation phase (Part 1).
Recommended Phase 2 dose (RP2D) of RP2 | 7 months
  RP2D of RP2 based on the safety and response data collected during the dose escalation phase (Part 1).

SECONDARY OUTCOMES:
Percentage of biologic activity | 20 weeks
  Percentage of subjects with biological activity determined by tumor biopsies and biomarker data
Percentage of subjects with detectable RP2 | 20 weeks
  Data gathered from blood, urine, swabs of injection site, dressings, and oral mucosa to determine the shedding and biodistribution of RP2.
Change in HSV-1 antibody levels | From Day 1 up to last dose (up to 4 months for dose escalation phase and up to 5.5 months for expansion phase)).
  Change in HSV-1 antibody levels during treatment compared to baseline
Percentage of overall response rate (ORR) | 3 years
  Percentage of ORR.
Median duration of response | 3 years
  Median duration of response of subjects
Median progression-free survival | 3 years
  Median duration of progression-free survival of subjects
Median overall survival | 3 years
  Median overall survival rate of subjects
Percentage of complete response (CR) | From Day 1 up to last dose (up to 8 weeks for escalation phase and up to 2 years for expansion phase).
  Percentage of subjects with a CR
Percentage of partial response (PR) | From Day 1 up to last dose (up to 8 weeks for escalation phase and up to 2 years for expansion phase).
  Percentage of subjects with a PR
Percentage of stable disease (SD) | From Day 1 up to last dose (up to 8 weeks for escalation phase and up to 2 years for expansion phase).
  Percentage of subjects with SD

CONTACTS AND LOCATIONS:
Overall Officials: Shaheen Kumar, MD, Study Director — Replimune Inc.
Locations (7):
- Spain (3):
  - Hospital Universitario d'Hebron, Barcelona
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Clinico de Valencia, Valencia
- United Kingdom (4):
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Bebington, Merseyside
  - The Royal Marsden NHS Foundation Trust, London
  - Churchill Hospital, Oxford
  - Royal Marsden Hospital, Sutton